CLINICAL TRIAL: NCT05043909
Title: Virtual Reality Training System on Oral Health Care for Dependency Elderly in Oral Hygiene Students: A Randomized Controlled Trial
Brief Title: The Effects of Virtual Reality and Augmented Reality Training System on Elderly Oral Care Skill for Oral Hygiene and Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KMUHIRB-SV(II)-20200071
Record Dates: First submitted 2021-08-27; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-08

CONDITIONS: Medical Education
Keywords: Dependency; Elderly; Medical Education; Oral Hygiene; Virtual Reality

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (EG) (Experimental): The students in EG received VR-based training for elderly oral health care at 2-week (Time 2), 4-week (Time 3), and 6-week (Time 4) follow-ups. The learning module was divided into three sessions according to the physical condition (1) Mild disability, (2) Semi-disability, (3) Total disability and oral condition, (1) wearing dentures, (2) missing teeth of the elderly. Students simulate the different physical and oral conditions of the elderly through virtual situations and provide suitable oral care methods. The whole training session took approximately two hours for each student; First, students were first given a short introduction to the VR system's use (10 minutes). Second, they were able to carry out oral care for the elderly while wearing VR goggles and using hand-controllers with the teaching and audio guides during the process (90 minutes), and an evaluation was taken after the intervention (20 minutes).
  Interventions: Behavioral: VR-based training
- Control Group (CG) (No Intervention): The students in CG do not receive any of the interventions. However, the same VR-based curriculum of oral health care on dependency elderly were provided at the end of the study.

INTERVENTIONS:
Behavioral: VR-based training — Students simulate the different physical and oral conditions of the elderly through virtual situations and provide suitable oral care methods. The whole training session took approximately two hours for each student; First, students were first given a short introduction to the VR system's use (10 minutes). Second, they were able to carry out oral care for the elderly while wearing VR goggles and using hand-controllers with the teaching and audio guides during the process (90 minutes), and an evaluation was taken after the intervention (20 minutes).
  Arms: Experimental Group (EG)

SUMMARY:
Virtual reality (VR) has been proposed as a promising technology for education since the combination of immersive and interactive features enables experiential learning. The study aimed to evaluate the effectiveness of VR-based training on oral health care for dependency elderly among oral hygiene students.

DETAILED DESCRIPTION:
A randomized controlled trial was conducted. Overall, the study recruited students from third grade of Department of Oral Hygiene students in Kaohsiung Medical University during 2021. The participants were randomly assigned to virtual-reality experimental (EG; n = 11) and control (CG; n = 12) groups. The students in EG received a 2-hour VR training for elderly oral health care at 2-week (Time 2), 4-week (Time 3) and 6-week (Time 4) follow-ups. Each student collected the data by a self-administrated questionnaire before and immediately after each of the intervention. Linear regression in generalized estimating equations (GEE) compare the differences between both groups.

ELIGIBILITY:
Inclusion Criteria:

* third grade of Department of Oral Hygiene students in Kaohsiung Medical University during the 2021 academic semester
* Participants have to take both the courses of 'Basic Medical Nursing Care' and 'Oral Health Care for Community People and Long-term Care Residents' before intervention.

Exclusion Criteria:

* none

Ages: 20 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Elderly oral care-related knowledge | Change from Baseline knowledge at 2-, 4-, 6-week follow-ups after the interventions
  Twenty items measured elderly oral care-related knowledge; for example, 'There is no need to consider the size of the interdental brush.' Possible responses included True (1), False (0), and I do not know (0), with possible scores ranged from 0 to 20; a higher score indicated a higher degree of oral-care-related knowledge. The KR-20 coefficient was 0.56 for this scale
Attitude toward elderly oral care | Change from Baseline attitude at 2-, 4-, 6-week follow-ups after the interventions
  Seven items measured attitude toward elderly oral care, for example, 'Assist disabled elderly to clean their teeth is annoying.' Each item was scored on a five-point Likert-type scale ranging from 1 (strongly disagree) to 5 (strongly agree). Possible scores ranged from 5 to 35; a higher score indicated a more positive attitude toward oral care for the elderly. Cronbach's alpha was 0.70 for this scale.
Self-efficacy of elderly oral care | Change from Baseline self-efficacy at 2-, 4-, 6-week follow-ups after the interventions
  Eleven items were used to evaluate the self-efficacy of elderly oral care. Students indicated their degrees of agreement with statements related to perceptions of personal ability concerning oral care for the elderly. For example, 'I am confident to remind disable elderly having regular dental visits every six months.' Each item was scored on a five-point Likert-type scale ranging from 1 (strongly disagree) to 5 (strongly agree). Possible scores ranged from 5 to 55; a higher score indicated more substantial confidence toward oral care for the elderly. Cronbach's alpha was 0.87 for this scale.
Intention to elderly oral care behaviors | Change from Baseline intentions at 2-, 4-, 6-week follow-ups after the interventions
  Twelve items were used to evaluate the intention to elderly oral care behavior for elderly. Students indicated their goals of adding new behaviors or modifying existing behaviors of oral care for the elderly. For example, 'I will take the initiative to assist disabled elderly to clean their dentures.' Each item was scored on a five-point Likert-type scale ranging from 1 (strongly disagree) to 5 (strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-Ling Huang, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, San Min District, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/09/NCT05043909/Prot_SAP_000.pdf